CLINICAL TRIAL: NCT05191797
Title: A Phase I/II Study of Bomedemstat Combined With Maintenance Immunotherapy for Patients With Newly Diagnosed Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Bomedemstat and Maintenance Immunotherapy for Treatment of Newly Diagnosed Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Rafael Santana-Davila, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122005; NCI-2021-13863 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA228944 (NIH); 10841 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Limited Stage Lung Small Cell Carcinoma
Keywords: Lung
MeSH Terms: interventions — bomedemstat; atezolizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bomedemstat, atezolizumab) (Experimental): Patients receive bomedemstat PO QD on days 1-21 and atezolizumab IV on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bomedemstat; Biological: Atezolizumab

INTERVENTIONS:
Drug: Bomedemstat — Given PO
  Other Names: 1990504-34-1; IMG 7289; IMG-7289; LSD-1 Inhibitor IMG-7289; Lysine-specific Demethylase 1 Inhibitor IMG-7289
Biological: Atezolizumab — Given IV
  Other Names: 1380723-44-3; Immunoglobulin G1; Anti-(human CD Antigen cd274) (Human Monoclonal MPDL3280A Heavy Chain); Disulfide with Human Monoclonal MPDL3280A Kappa-chain; Dimer; MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq

SUMMARY:
This phase I/II trial studies the side effects of bomedemstat and maintenance immunotherapy with atezolizumab and to see how well they work in treating patients with newly diagnosed extensive stage small cell lung cancer. Bomedemstat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving bomedemstat and atezolizumab may work better in treating patients with extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive bomedemstat orally (PO) once daily (QD) on days 1-21 and atezolizumab intravenously (IV) on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or older and willing and able to provide written informed consent
* Histologically confirmed diagnosis of extensive stage small-cell lung cancer (ES-SCLC)

  * Note: Previously treated limited stage SCLC (LS-SCLC) patients are eligible if disease progression had occurred following completion of definitive treatment for LS-SCLC. Determination of disease progression after prior therapy for LS-SCLC is at the discretion of the investigator
* Having received four cycles of platinum-etoposide concurrent with three or four cycles of immune checkpoint inhibitor as induction systemic therapy for ES-SCLC immediately prior to study enrollment (see below for definitions). Note that immune checkpoint inhibitor may have been omitted from the first cycle only

  * Platinum is defined as cisplatin or carboplatin. Immune checkpoint inhibitor is defined as atezolizumab, durvalumab, or other anti-PDL1 or anti-PD1 monoclonal antibody that is approved by the United States (US) Food and Drug Administration for first-line treatment of ES-SCLC in combination with platinum and etoposide at the time of treatment receipt. Immediately prior is defined as receipt of cycle 1 day 1 of platinum-etoposide +/- immune checkpoint inhibitor no more than 112 days prior to cycle 1 day 1 of study treatment, and administration of fourth cycle of platinum-etoposide and immune checkpoint inhibitor no more than 30 days prior to cycle 1 day 1 of study treatment
* Eligible to receive maintenance atezolizumab, as defined by stable disease or better, following induction platinum-etoposide and immune checkpoint inhibitor. Determination of response to induction therapy is at the discretion of the investigator. Investigators should contact the principal investigator (PI) if clarification is needed
* Eastern Cooperative Oncology Group (ECOG performance status of =< 2)
* Minimum life expectancy of >= 12 weeks

  * Note: myeloid growth factor use within 14 days of study treatment initiation is not permitted. Growth factor may have been previously administered during induction chemoimmunotherapy
* Platelet count (Plt) >= 75 x 10^3/mcL (without transfusion)
* Hemoglobin (Hgb) >= 8.0 g/dL (transfusion is permitted)
* Calculated glomerular filtration rate (GFR; using the Cockcroft-Gault equation) >= 40 mL/min or serum creatinine =< 1.5 x upper limit of normal
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) or =< 3 x ULN for subjects with Gilbert's disease
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN if evidence of hepatic involvement by malignant disease)
* International normalized ratio (INR) < 1.5 x upper limit of normal (only in patients not receiving anticoagulant agents at baseline)

  * Note: there is no INR or activated partial thromboplastin time (aPTT) threshold for patients who are receiving anticoagulant agents at baseline, but patients must be on a stable dose of anticoagulant, and discontinuation of all anticoagulation while the platelet count is below 50 x 10^3/mcL must be deemed appropriate for the patient by the investigator prior to enrollment
* Activated partial thromboplastin time (aPTT) < 1.5 x the local upper limit of normal (only in patients not receiving anticoagulant agents at baseline)

  * Note: there is no INR or aPTT threshold for patients who are receiving anticoagulant agents at baseline, but patients must be on a stable dose of anticoagulant, and discontinuation of all anticoagulation while the platelet count is below 50 x 10^3/mcL must be deemed appropriate for the patient by the investigator prior to enrollment
* Able to swallow capsules
* Amenable to peripheral blood sampling during the study
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 28 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects who are sexually active with female partner(s) of childbearing potential should be willing to use an adequate method of contraception starting with the first dose of study therapy through 28 days after the last dose of study therapy

Exclusion Criteria:

* Prior receipt of systemic therapy for ES-SCLC other than four cycles of induction platinum-etoposide and immune checkpoint inhibitor
* Diagnosis of LS-SCLC that has not been previously treated
* Receipt of radiation therapy for symptomatic deterioration and/or radiographic disease progression that was administered after initiation of induction platinum-etoposide and immune checkpoint inhibitor. Note: the presence of untreated asymptomatic brain metastasis, or a history of receipt of radiation to brain metastasis that was not initiated in response to symptomatic deterioration and/or radiographic disease progression following initiation of induction systemic therapy, does not preclude study participation. Investigators should contact the PI if clarification is needed
* Anticipated use of prophylactic cranial irradiation or consolidative thoracic radiation therapy during study participation. Note: Palliative radiation to the central nervous system (CNS) for new CNS disease that develops during study participation is allowed
* History of prior immune-related adverse event or other toxicity associated with immune checkpoint inhibitor that precludes safe administration of maintenance atezolizumab, in the opinion of the investigator
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at doses not to exceed 10 mg/d of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Active autoimmune disease requiring systemic immunosuppression or history of autoimmune disease requiring systemic immunosuppression within the last 2 years

  * Note: Systemic immunosuppression should be interpreted as systemic glucocorticoids at a dose of greater than 10 mg/day of prednisone or equivalent, systemic biologic agents including monoclonal antibodies against inflammatory mediators, or small molecule agents. Investigators should contact the PI if clarification is needed
* Active pneumonitis or interstitial lung disease (ILD), or a history of pneumonitis/ILD, which required systemic immunosuppression (e.g. corticosteroids)
* Known bleeding disorder (e.g., dysfibrinogenaemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation [DIC], fibrinogen deficiency, or other clotting factor deficiency), at the discretion of the investigator
* History of severe thrombocytopenia or platelet dysfunction (e.g. immune thrombocytopenic purpura), at the discretion of the investigator
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to bomedemstat or LSD1 inhibitors (i.e., monoamine oxidase inhibitors; MAOIs) that contraindicates their participation
* Any hypersensitivity to PD-1/PD-L1 targeting agents
* Current use of monoamine oxidase A and B inhibitors (MAOIs)
* Current use of a prohibited medication (e.g. romiplostim) or expected to require any of these medications during treatment with the investigational drug
* Current or anticipated use of an antiplatelet (e.g. clopidogrel), anticoagulant (e.g. warfarin or apixaban), or nonsteroidal anti-inflammatory drug (NSAID) with antiplatelet activity (e.g. aspirin, ibuprofen), that, in the opinion of the investigator, could NOT be safely discontinued when the subject's platelet count decreases below 50 x 10^3/mcL
* Has undergone major surgery within 4 weeks prior to starting study drug and/or has not recovered from side effects of such surgery. Note: Major surgery and recovery are defined at the discretion of the investigator
* Receipt of a live vaccine within 30 days of first dose of study therapy
* Uncontrolled active infection
* Any concomitant active malignancy considered clinically significant by the investigator
* Known human immunodeficiency virus (HIV) infection or known active hepatitis B or hepatitis C virus infection (testing will not be conducted as part of screening procedures)
* History of any illness/impairment of gastrointestinal (GI) function that might interfere with drug absorption (e.g. chronic diarrhea), confound the study results or pose an additional risk to the patient by participation in the study
* Use of an investigational agent within 28 days, or the equivalent of at least 7 half-lives of that agent, whichever is the shorter, prior to the study day 1
* Females who are pregnant or breastfeeding or plan to become pregnant or breastfeed at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Santana-Davila, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: Years] | 63 [58 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity (DLT)
Description: DLT to bomedemstat combined with atezolizumab is defined as the occurrence of any of the following toxicities by CTCAE 5.03 determined to be possibly, probably, or likely related to bomedemstat or atezolizumab occurring within 21 days of initiation of treatment. The specific events are:
  - Grade 4 non-hematologic toxicity (not laboratory).
  * Grade 3 non-hematologic toxicity (not laboratory) lasting >3 days despite optimal supportive care.
  * Any Grade 3 or Grade 4 non-hematologic laboratory value if:
    * Medical intervention is required to treat the patient, or
    * The abnormality leads to hospitalization
    * Thrombocytopenia leading to clinically significant sequelae (i.e., a clinically significant bleeding event or the need for prophylactic transfusions).
    * Febrile neutropenia.
    * Grade 5 toxicity.
Time Frame: Up to 21 days from initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Progression Free Survival
Description: Distributions for time-to-event outcomes will be evaluated using the method of Kaplan-Meier. For point estimates at landmark times, the associated 95% confidence interval (CI) will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function.
Time Frame: From the date of study enrollment up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Number analyzed (Participants) | 3
months | 3.82 [1.53 to 6.11]

3. Primary Outcome: Incidence Patients Experiencing Adverse Events
Description: Only adverse events that meet the following definition will be recorded:
  1. All grade 3 and higher adverse events
  2. Grade 1-2 adverse events that require medical intervention, i.e. initiation of a new medication, or are otherwise clinically significant at the discretion of the investigator
  3. Any adverse event that requires a dose reduction or dose delay of either bomedemstat or atezolizumab Adverse events will be recorded from Cycle 1 Day 1 until the Safety Monitoring visit performed according to the Study Calendar (Section 7.0), using the Adverse Event case report forms/worksheets. For subjects who discontinue study therapy for a reason other than disease progression and are being followed with Monitoring visits (Section 8.5.3.3), adverse events should continue to be monitored. Adverse events related to either bomedemstat or atezolizumab will be followed until resolution or stabilization of the AE or until the beginning of a new anti-neoplastic therapy, whichever occurs first.
Time Frame: From initial of treatment, up to 30 days after discontinuation of study treatment, up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Number analyzed (Participants) | 3
Participants
  Elevated Creatinine | 1
  Transaminitis | 1
  Syncope | 1
  H. Pylori | 1
  Fatigue | 1
  Shingles | 1
  Maculopapular Rash | 1
  Left Lower Extremity Pain | 1
  Left Lower Extremity Weaskness | 1

4. Secondary Outcome: Overall Survival
Description: Distributions for time-to-event outcomes will be evaluated using the method of Kaplan-Meier. For point estimates at landmark times, the associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function.
Time Frame: From the date of study enrollment until death from any cause up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
Number analyzed (Participants) | 3
Months | 15.1 [6.56 to 23.64]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored for up to 2 years; serious and/or other adverse events were assessed up to 1 year, 3 months
Description: Only adverse events that meet the following definition will be recorded:
  All grade 3 and higher adverse events Grade 1-2 adverse events that require medical intervention or are otherwise clinically significant at the discretion of the investigator Any adverse event that requires a dose reduction or dose delay of either bomedemstat or atezolizumab Adverse events will be recorded from Cycle 1 Day 1 until 30 days post EOT.
Arm/Group | Treatment (Bomedemstat, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bomedemstat, Atezolizumab) (N=3)
Elevated Creatinine (Investigations) | 1 (1)
Transaminitis (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
H. Pylori (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Left Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Lower Extremity Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05191797/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05191797/ICF_000.pdf